CLINICAL TRIAL: NCT03594721
Title: Clinical Trial Evaluation of a Test Serum Post HEV (High Energy Visible) Light Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKM18-MARV-HEV
Record Dates: First submitted 2018-06-25; First posted 2018-07-20 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Blue Light Damage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitzpatrick Skin Types I-III (Experimental): Volunteers will return to the clinic after Baseline for 10 additional, consecutive days for study staff to apply approximately 2 mg/cm2 or 50 µL of test product to the appropriate 5x5cm2 test location on the lower back. Volunteers will have digital images of the three (3) areas on the lower back that comprise the entire test region taken at Baseline, and 24hrs post 90J/cm2 HEV light exposure.
  Interventions: Other: Marvel AM
- Fitzpatrick Skin Types IV-V (Experimental): Volunteers will return to the clinic after Baseline for 10 additional, consecutive days for study staff to apply approximately 2 mg/cm2 or 50 µL of test product to the appropriate 5x5cm2 test location on the lower back. Volunteers will have digital images of the three (3) areas on the lower back that comprise the entire test region taken at Baseline, and 24hrs post 90J/cm2 HEV light exposure.
  Interventions: Other: Marvel AM

INTERVENTIONS:
Other: Marvel AM — Study staff will perform each application of approximately 2 mg/cm2 or 50 µL of test product to the appropriate 5x5cm2 test location on the lower back at each of ten sequential visits.

SUMMARY:
To evaluate 10 days of pretreatment with a serum (Test Product/Marvel AM) to the lower back, followed by a single exposure of 90J/cm2 HEV (High Energy Visible) light {400-450nm wavelengths} in healthy male or female volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers can be male or female, 18 to 65 years of age with no known medical conditions that, in the investigator's opinion, may interfere with study participation.
* Volunteers must sign a written informed consent.
* Volunteers must fall within Fitzpatrick Skin Type I-V.
* Volunteers must be willing to avoid sun exposure to the study treatment area (lower back) for the duration of the study.
* Volunteers must commit to meeting all study requirements, including 11 days of sequential office visits for product application, HEV exposure, biopsy and suture removal.

Exclusion Criteria:

* Volunteers who are pregnant, breast feeding or planning a pregnancy during the study period.
* Have used within the month before inclusion, any systemic medication for more than 5 consecutive days (e.g. steroidal and non-steroidal anti-inflammatory drugs, insulin, antihistamines, antihypertensive, antibiotics-e.g quinolone, tetracycline, thiazides, fluoroquinolones), or any medication known to cause abnormal responses to HEV light exposure (e.g. vitamin A derivatives, psoralen, aminolevulinic acid derivatives, etc.), or having planned to use these medications during the study.
* Volunteers who have damaged skin in close proximity to test sites (e.g. sunburn, uneven skin tones, tattoos, scars or other disfigurations)
* Volunteers who have used a prescription hydroquinone, non-hydroquinone skin lightening or brightening agent, or like product in the test area, within the past 3 months.
* Volunteers who have used a non-prescription cosmetic anti-aging or skin lightening product known to affect dyschromia or hyperpigmentation, in the test area, within the past 4 weeks.
* Volunteers who have a history of scarring, hypertrophic scarring or keloid formation anywhere on their body.
* Volunteers with a known sensitivity to lidocaine or epinephrine.
* Volunteers who are unwilling or unable to comply with the requirements of the protocol, including ability to complete all study visits within the proscribed study visit window for any reason(s).
* Volunteers with any disorder that may prevent compliance, such as history of chronic alcohol or drug abuse, significant mental or nervous disorder or other illness that would, in the evaluator's opinion, interfere with the study.
* Have participated, or are participating in, another study within the past 4 weeks.
* Any dermatologic disorder which, in the investigator's opinion, may interfere with the accurate evaluation of the study treatment area (lower back), but not limited to melasma, any active inflammatory skin condition (i.e. post inflammatory hyperpigmentation), severe acne vulgaris, acne conglobata, acne fulminans, seborrheic dermatitis, and lupus erythematosus.
* Volunteers who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study products.
* Concurrent therapy with any medication either topical or oral which, in the investigator's opinion, may interfere with evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Photographs for detection of changes in the treatment areas. | Baseline, Day 11
  Photographic images of the lower back, will be captured utilizing a digital system. Photos may be taken from multiple angles to allow for easy detection of changes in the treatment areas.
Chromamemter instrument will be used to assess the change of color on the skin. | Baseline, Day 11
  Chromameter instrument will be used to measure color on the skin.
Punch biopsies will be taken from the 3 different areas on the lower back to evaluate histological changes. | Baseline, Day 11
  Punch biopsies will be taken from the 3 different areas on the lower back for histological evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Makino, Study Director — Allergan
Locations (1):
- McDaniel Institute of Anti Aging Research, Virginia Beach, Virginia, United States

IPD SHARING:
Plan to Share IPD: No